CLINICAL TRIAL: NCT01542450
Title: A Randomised, Open-labelled, Single-centre, Two-period Crossover Trial Investigating the Pharmacodynamics and Pharmacokinetics of Single s.c. Doses of NN304 (Insulin Detemir) and NPH Human Insulin in Japanese Subjects With Type 1 Diabetes Mellitus
Brief Title: Pharmacokinetics of Insulin Detemir in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1475; JapicCTI-R070015 (Registry Identifier: JAPIC)
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin NPH
- Treatment period 2 (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Single dose of 0.3 U/kg administered subcutaneously (s.c. under the skin) in each treatment period separated by a washout period of 4-28 days
Drug: insulin NPH — Single dose of 0.3 U/kg administered subcutaneously (s.c. under the skin) in each treatment period separated by a washout period of 4-28 days

SUMMARY:
This trial is conducted in Japan. The aim for this trial is to investigate the pharmacodynamics and pharmacokinetics of insulin detemir and insulin NPH in Japanese subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* HbA1c (glycosylated haemoglobin) maximum 9.0%
* Duration of diabetes at least 1 year
* Body Mass Index (BMI) maximum 25.0 kg/m^2

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Proliferative retinopathy or maculopathy requiring acute treatment as judged by the Investigator
* Impaired hepatic function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated / untreated hypertension
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies, positive
* Known or suspected allergy against the trial products or related products including the components
* Previous history of serious allergy or anaphylactic reaction
* Any disease or condition which the Investigator feel would interfere with the trial participation or evaluation of the results
* Severe late-phase diabetic complications including nephropathy
* Blood donation of more than 400 mL (inclusive) in total within the last 12 weeks or more than 200 mL (inclusive) in total within the last 3 weeks
* Known or suspected alcohol and illicit substance abuse or dependence
* Pregnancy, breast-feeding (within a year after labour) or the intention to become pregnant
* The receipt of any investigational drug within the last 12 weeks prior to this trial
* Current or anticipated treatment with systemic corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The ratio of area under the glucose infusion rate curve (AUCGIR) 0-5 hours to AUCGIR 0-24 hours

SECONDARY OUTCOMES:
AUCGIR, area under the glucose infusion rate value curve
GIRmax, the maximum GIR value
tmax GIR, time to maximum GIR value
Cmax, maximum concentration
Area under the curve
tmax, time to maximum concentration
MRT, mean residence time
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Irie S, Matsumura Y, Hirano K. Pharmacokinetics and Pharmacodynamics of Single Dose Insulin Detemir, Long-acting soluble insulin analogue compared to NPH insulin in Patients with type 1 Diabetes Mellitus. Journal of Clinical Ther. and Med. 2007; 5 (23): 349-356
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com